CLINICAL TRIAL: NCT06138275
Title: A Phase 2 Study of Elranatamab as Consolidation After Idecabtagene Vicleucel in Relapsed Refractory Multiple Myeloma
Brief Title: Elranatamab in R/R Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Noopur Raje, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-402
Record Dates: First submitted 2023-10-28; First posted 2023-11-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Refractory Multiple Myeloma; Relapse Multiple Myeloma; Multiple Myeloma
Keywords: relapsed/refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elranatamab (Experimental): Elranatamab subcutaneous injections at pre-determined doses, administered at the following timepoints during each 28-day cycle: Cycle 1: Days 1, 4, 8, 15, and 22; Cycle 2: Days 1, 8, 15, and 22 ; Cycles 3-6: Days 1 and 15
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — subcutaneous (under the skin) injection

SUMMARY:
This research is being done to see if the study drug, elranatamab, reduces the risk of disease progression (worsening disease) after idecabtagene vicleucel in relapsed refractory multiple myeloma.

DETAILED DESCRIPTION:
This is an open label phase II study that will enroll patients with relapsed and refractory multiple myeloma after four or more lines of therapy who received idecabtagene vicleucel as standard of care.

The research involves study visits and receiving the study drug. Participants will receive the study drug, elranatamab, for up to 6 months and will be followed for as long as they remain in the study, until confirmed progressive disease (disease worsening), or until initiation of other myeloma treatment.

Elranatamab is a type of antibody (a protein produced by the body's immune system when it detects harmful substances) that works by binding to both T-cells (part of the immune system) and myeloma cells. The drug then activates T-cells to kill the myeloma cells. In this study we are researching whether multiple myeloma progresses after elranatamab administration. The U.S. Food and Drug Administration (FDA) has not approved elranatamab as a treatment for any disease.

It is expected that about 32 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participant has given voluntary signed written informed consent before performance of any study related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to their future medical care.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Male or female participants age ≥ 18 years
* The effects of elranatamab on the developing human fetus are unknown. For this reason and because anti-BCMA bispecific antibodies are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of elranatamab administration.
* Prior diagnosis of MM as defined according to IMWG criteria.
* Measurable disease of multiple myeloma as defined by at least one of the following prior to idecabtagene vicleucel infusion:

  * Serum monoclonal protein ≥ 0.5 g/dL. Patients with IgD disease and lower amounts of monoclonal protein may be permitted to enroll with PI approval
  * ≥ 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum free light chain ≥ 100 mg/L (10 mg/dL) and abnormal serum free kappa to serum free kappa light chain ratio (<0.26 or >1.65)
* Previously treated relapsed and refractory multiple myeloma following idecabtagene vicleucel as infusion as standard of care who have achieved at least a PR or better per IMWG criteria. Patients will have received idecabtagene per label including after at least 4 prior lines of therapy and relapsed after an immunomodulatory drug (IMiD), a proteasome inhibitor and an Anti-CD38 monoclonal antibody
* left ventricular ejection fraction (LVEF) ≥40% as determined by a multiple gated acquisition scan (MUGA) scan or echocardiogram (ECHO).
* Participants must meet the following organ and marrow function as defined below:

  * Absolute neutrophil count ≥1000/microlitre (mcL). Use of granulocyte-colony stimulating factors is permitted if completed at least 7 days prior to planned start of dosing.
  * Platelet count ≥25,000/mcL. Platelet transfusion support is permitted if completed at least 7 days prior to planned start of dosing.
  * Hemoglobin ≥8 g/dL. Red blood cell transfusion support is permitted if completed at least 7 days prior to planned start of dosing.
  * Calculated creatinine clearance ≥30 mL/min by Cockcroft-Gault equation.
  * Patient has adequate hepatic function, as evidenced by each of the following:

    * Serum total bilirubin <2 mg/dL; and
    * Serum aspartate transaminase (ALT) and/or aspartate transaminase (AST) values < 2.5 × the upper limit of normal (ULN) of the institutional laboratory reference range. Patients with elevated bilirubin due to Gilbert's syndrome may be permitted with PI approval (e.g. total bilirubin <3 mg/dL and normal direct bilirubin).
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria:

* Patients with smoldering MM, plasma cell leukemia, POEMS syndrome, or amyloidosis are excluded from this trial.
* Stem cell transplant within 12 weeks prior to enrollment or active graft-versus-host disease (GVHD).
* Active hepatitis B virus, hepatitis C virus, Severe acute respiratory syndrome coronavirus 2 (SARS-CoV2), HIV, or any active, uncontrolled bacterial, fungal, or viral infection. Active infections must be resolved at least 14 days prior to enrollment.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, defined as any of the following within 6 months prior to enrollment:

  * Acute myocardial infarction or acute coronary syndromes (eg, unstable angina, coronary artery bypass graft, coronary angioplasty or stenting, symptomatic pericardial effusion);
  * Clinically significant cardiac arrhythmias (eg, uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
  * Thromboembolic or cerebrovascular events (eg, transient ischemic attack, cerebrovascular accident, deep vein thrombosis [unless associated with a central venous access complication] or pulmonary embolism);
  * Prolonged QT syndrome (or triplicate average QTcF >470 msec at screening).
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
* Ongoing Grade ≥2 peripheral sensory or motor neuropathy.
* History of Guillain-Barré syndrome (GBS) or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.
* Previous treatment with an anti-BCMA (B-cell maturation antigen) bispecific antibody.
* Pregnant women are excluded from this study because elranatamab is an anti-BCMA bispecific antibody agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with elranatamab, breastfeeding should be discontinued if the mother is treated with elranatamab.

Known or suspected hypersensitivity to the study intervention or any of its excipients.

Participants who are receiving any other investigational agents for this condition (if appropriate only).

Live attenuated vaccine must not be administered within 4 weeks of the first dose of study intervention.

Toxicity from previous anticancer therapy must resolve to baseline levels or to grade ≤1, except for alopecia and peripheral neuropathy.

Other surgical (including major surgery within 14 days prior to enrollment), medical or psychiatric conditions including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate or stringent CR (sCR) post consolidation therapy | The time from start of treatment to first date that progressive disease is objectively documented or death due to any cause, for up to 5 years. Participants without events reported are censored at the last disease evaluation.
  Disease response will be assessed using the International Myeloma Working Group Response Criteria (IMWG)
Progression-free survival | The time from registration to the earlier of progression or death due to any cause, for up to 5 years. Participants alive without disease progression are censored at date of last disease evaluation
  Progression-Free Survival (PFS) is defined as the time from or registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. This will be estimated with the Kaplan-Meier method and summarized with medians and 95% confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 3 years
  Adverse events will be evaluated using CTCAE version 5
Objective response rate (ORR) | From start of treatment to 2 years post-treatment
  ORR will be evaluated using the IMWG Uniform Response criteria
Overall survival (OS) | From start of treatment to 2 years post-treatment
  Overall Survival (OS) is defined as the time from or registration to death due to any cause, or censored at date last known alive. Estimated with the Kaplan-Meier method and summarized with medians and 95% confidence intervals.
Minimum Residual Disease (MRD)-positive to MRD-negative conversion rate | 6 months
  MRD-positive to MRD-negative conversion rate is the proportion of MRD-positive participants that become MRD-negative. Point estimates of MRD positivity and negativity rates will be calculated along with the 2-sided 95% CIs using the Clopper-Pearson method.
Rate of sustained MRD-negativity of ≥6 or ≥12 months | 6 years
  Sustained MRD negativity rate is the proportion of participants with MRD negativity sustained over at least 6 months or at least 12 months from the date of first dose until the first documentation of confirmed PD, death or start of new anticancer therapy. Point estimates of MRD negativity rate will be calculated along with the 2-sided 95% Confidence Interval (CIs) using the Clopper-Pearson method.
Time to MRD-negativity | From start of treatment to 2 years post-treatment
  MRD negativity rate is the proportion of participants with negative MRD per IMWG sequencing criteria from the date of first dose until the first documentation of confirmed PD, death or start of new anticancer therapy. Point estimates of MRD negativity rate will be calculated along with the 2-sided 95% CIs using the Clopper-Pearson method.
Duration of response (DOR) | From start of treatment to 2 years post-treatment
  The following description information was pulled from NIH: Duration of response is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response. This is estimated with the Kaplan-Meier method and summarized with medians and 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation